CLINICAL TRIAL: NCT06874569
Title: Assistant Professor and the Principle Investigator
Brief Title: A Comparing Transversalis Fascia Plane Block and Quadratus Lumborum Block for Post-Cesarean Pain Management: Efficacy, Execution Time, and Practicality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Collaborators: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Ayman Mohamady Eldemrdash, Principal Investigator, Aswan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: regional block post C-section
Record Dates: First submitted 2025-02-12; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Regional Anesthesia Block

STUDY DESIGN:
Intervention Model Description: Participants were randomized into three equal groups (n = 36 per group) to receive either Transversus Abdominis Plane Block (TAPB, control), Transversalis Fascia Plane Block (TFPB), or Quadratus Lumborum Block (QLB). A computer-generated randomization sequence was used, and group allocations were concealed in sealed opaque envelopes, which were opened only after enrollment. Although the anesthesiologist performing the block knew the group allocation, patients and outcome assessors were blinded to minimize bias.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: A computer-generated randomization sequence was used, and group allocations were concealed in sealed opaque envelopes, which were opened only after enrollment. Although the anesthesiologist performing the block knew the group allocation, patients and outcome assessors were blinded to minimize bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TAP Block (Active Comparator): TAP Block: A linear high-frequency probe (6-13 MHz) was placed transversely along the midaxillary line to visualize the external oblique, internal oblique, and transversus abdominis muscles. Using an in-plane approach, a 21G SonoPlex, STIM (PAJUNK, Germany), was advanced, and after hydro-dissection with 1-2 mL saline, 20 mL of 0.25% bupivacaine (Marcaine, AstraZeneca, Sweden) was injected into the plane between the internal oblique and transversus abdominis muscles.
  Interventions: Procedure: TAP Block:
- TFP Block (Experimental): TFP Block: With a linear probe, the transversalis fascia was identified between the internal oblique and transversus abdominis muscles. An in-plane technique was used to insert a 21G needle, and following confirmation of correct placement with hydro-dissection, 20 mL of 0.25% bupivacaine was administered bilaterally.
  Interventions: Procedure: TFP Block:
- QLB: (Experimental): QLB: A low-frequency curvilinear probe (2-5 MHz) was used to identify the quadratus lumborum muscle and adjacent structures. The needle was advanced in-plane until it reached the targeted region adjacent to the quadratus lumborum, where after hydro-dissection, 20 mL of 0.25% bupivacaine was injected bilaterally.
  Interventions: Procedure: QLB:

INTERVENTIONS:
Procedure: TAP Block: — TAP Block: A linear high-frequency probe (6-13 MHz) was placed transversely along the midaxillary line to visualize the external oblique, internal oblique, and transversus abdominis muscles. Using an in-plane approach, a 21G SonoPlex, STIM (PAJUNK, Germany), was advanced, and after hydro-dissection with 1-2 mL saline, 20 mL of 0.25% bupivacaine (Marcaine, AstraZeneca, Sweden) was injected into the plane between the internal oblique and transversus abdominis muscles.
  Arms: TAP Block
Procedure: TFP Block: — TFP Block: With a linear probe, the transversalis fascia was identified between the internal oblique and transversus abdominis muscles. An in-plane technique was used to insert a 21G needle, and following confirmation of correct placement with hydro-dissection, 20 mL of 0.25% bupivacaine was administered bilaterally.
  Arms: TFP Block
Procedure: QLB: — QLB: A low-frequency curvilinear probe (2-5 MHz) was used to identify the quadratus lumborum muscle and adjacent structures. The needle was advanced in-plane until it reached the targeted region adjacent to the quadratus lumborum, where after hydro-dissection, 20 mL of 0.25% bupivacaine was injected bilaterally.
  Arms: QLB:

SUMMARY:
Transversalis Fascia Plane Block (TFPB) and Quadratus Lumborum Block (QLB) provide superior analgesia to Transversus Abdominis Plane Block (TAPB) for post-cesarean pain management. This study evaluates whether TFPB or QLB is preferable when their analgesic efficacy is nearly equal, focusing on ease of performance and execution time.

DETAILED DESCRIPTION:
Cesarean delivery is one of the most common surgical procedures worldwide and is associated with significant postoperative pain that includes both somatic and visceral components . Effective pain management not only enhances patient comfort and satisfaction but also facilitates early mobilization and reduces maternal morbidity . Although the Transversus Abdominis Plane (TAP) block is widely used as part of a multimodal analgesia strategy, its relatively short duration of action and limited ability to relieve visceral pain have prompted the search for improved alternatives .

Recent advancements in ultrasound-guided regional anesthesia have introduced the Quadratus Lumborum Block (QLB) and the Transversalis Fascia Plane Block (TFPB) as promising techniques for post-cesarean analgesia. The QLB, first described by Blanco (2007) , offers extended analgesia due to its paravertebral spread, thereby addressing both somatic and visceral pain . In contrast, TFPB targets the transversalis fascia to block the T12 and L1 nerves, effectively reducing postoperative pain following cesarean delivery . Although both QLB and TFPB have been shown to provide superior analgesia compared to TAP blocks , limited data exist regarding their comparative ease of performance and procedural efficiency.

Given that the analgesic efficacy of TFPB and QLB appears comparable, it is essential to evaluate additional factors such as the time required to perform the block and the technical ease of the procedure. These factors are particularly critical in high-volume obstetric settings, where efficiency can significantly impact clinical workflow . Therefore, this study aims to compare TFPB and QLB not only in terms of analgesic efficacy but also regarding ease of performance and execution time, to determine which technique may be preferable for post-cesarean analgesia.

ELIGIBILITY:
Inclusion Criteria:-

1. Pregnant women aged 20-40 years scheduled for elective cesarean delivery under spinal anesthesia .
2. American Society of Anesthesiologists (ASA) physical status of II
3. Body mass index (BMI) of less than 35 kg/m² .

Exclusion criteria :-

1. History of allergy to local anesthetics.
2. Contraindications to regional anesthesia (such as coagulopathy or infection at the injection site).
3. Severe systemic diseases (renal, hepatic, or cardiovascular dysfunction).
4. weight less than 50 kg (to avoid exceeding safe doses of local anesthetic).
5. pregnancy complications like severe preeclampsia, eclampsia, or postpartum hemorrhage.

   -

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 108 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
postoperative pain by Numeric Pain Rating Scale | 6 ,12 and 24 hours
  The primary outcome, postoperative pain, was assessed using the Numeric Pain Rating Scale (NRS) at predefined intervals: 6, 12, and 24 hours postoperatively. Pain scores were documented by trained nursing staff blinded to the intervention. Opioid administration was standardized-patients received nalbuphine in 2 mg increments as needed (NRS more than 4), with a maximum dose of 10 mg in 24 hours.Minimum score 0 (no pain) and maximum 10 (severe pain). The lower the number the more free pain and the more high scale the more pain present.

CONTACTS AND LOCATIONS:
Locations (1):
- Ayman Mohamady Eldemrdash, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferguson JE, Tubog TD, Johnson W, Evans H, Furstein J. Quadratus Lumborum Block and Transversus Abdominis Plane Block in Non-emergency Cesarean Delivery: A Systematic Review and Meta-analysis. J Perianesth Nurs. 2024 Apr;39(2):226-234. doi: 10.1016/j.jopan.2023.07.017. Epub 2023 Oct 20. PMID 37865903
- [Background] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488
- [Background] Benedicta R, Jain MK, Dixit N, Shivappagoudar VM. The Efficacy of Ultrasound-guided Transversus Abdominis Plane Block Versus Quadratus Lumborum Block for Postoperative Analgesia in Lower-Segment Cesarean Section with Low-Dose Bupivacaine: A Randomized Controlled Trial. Anesth Essays Res. 2022 Apr-Jun;16(2):203-207. doi: 10.4103/aer.aer_84_22. Epub 2022 Sep 6. PMID 36447913
- See also: https://pubmed.ncbi.nlm.nih.gov/36447913/ — https://pubmed.ncbi.nlm.nih.gov/36447913/